CLINICAL TRIAL: NCT03904745
Title: Effect of Oxytocin Antagonists on Implantation Success Rates of Frozen-thawed Embryo Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Atosiban study
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Infertility, Female
Keywords: in vitro fertilization; atosiban; embryo transfer; oxytocin antagonist
MeSH Terms: conditions — Infertility, Female | interventions — atosiban

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atosiban used before embryo transfer (Experimental): the patients in this group will be administered 6,75mg atosiban intravenously.
  Interventions: Drug: Atosiban
- Control group (No Intervention): the patients in this group will not be administered atosiban before embryo transfer.

INTERVENTIONS:
Drug: Atosiban — 6,75mg of atosiban will be administered intravenously 30 minutes before embryo transfer
  Arms: Atosiban used before embryo transfer

SUMMARY:
Uterine contraction has a negative impact on implantation and pregnancy rates. Inhibition of oxytocin receptors decreases uterine contraction frequency both on pregnant and non-pregnant women. Atosiban has been studied as an oxytocin antagonist to decrease uterine contraction frequency in order to increase implantation and pregnancy rates in assisted reproduction. Previous studies have studied 37,5mg total dose which was used both before and during embryo transfer, and found atosiban to be effective in increasing implantation and pregnancy rates. We aim to use a single dose of 6,75mg atosiban before embryo transfer, in order to decrease the dose and cost and possibly introduce a simpler protocol. Our study will also be the first randomized clinical study which investigates the effect of atosiban on frozen-thawed embryo transfer cycles.

DETAILED DESCRIPTION:
Inhibition of uterine contractions in order to increase implantation rates have been studied on several agents in the last two decades. Beta-adrenergic agonists and non-steroidal anti-inflammatory drugs have been shown to have no benefit on implantation rates. Vasopressin V1a and oxytocin receptor antagonist atosiban was first studied on premature labor patients and found to be effective.

Endometrium-originated oxytocin can possibly stimulate myometrium and have a negative impact on embryo implantation. Inhibition of oxytocin receptors has been shown to reduce uterine contraction frequency in non-pregnant women. Atosiban has been studied on assisted reproductive technologies in the last decade and has been shown to be effective on increasing implantation and clinical pregnancy rates. However, previous studies have used a 37,5 mg total dose of atosiban which was used both before and during embryo transfer. We aim to use a single and low dose of 6,75mg atosiban only before embryo transfer, which is simpler and cheaper and the medication given to patient is significantly lower. If we can demostrate the positive effect of our protocol, it can be suggested to be used routinely in all in vitro fertilization cycles. Additionally, our study is an original study in terms of being the first randomized clinical trial studying the effect of atosiban on frozen-thawed embryo transfer cycles.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women applied to assisted reproduction clinic
* Follicle stimulating hormone < 12
* Body mass index < 25
* Patients whom antagonist protocol will be used
* Patients whom at least 2 good-quality embryos obtained
* Patients who are volunteer

Exclusion Criteria:

* Severe male factor (Sperm concentration <5 M/ml, progressive sperm motility <%10)
* Uterine anomaly
* Hydrosalphynx
* Difficult embryo transfer
* Patients who previously had a diagnosis of endometriosis and / or adenomyosis
* Endocrine problems (hypothyroidism, hyperthyroidism, hyperprolactinemia, premature ovarian insufficiency)
* Having more than 3 in vitro fertilization failure
* Refusing to participate

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-12-21 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rates | 1 year
  Pregnancy rates of the participants

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bezmialem University, Istanbul
  - Yeditepe University, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bossmar T, Akerlund M, Fantoni G, Szamatowicz J, Melin P, Maggi M. Receptors for and myometrial responses to oxytocin and vasopressin in preterm and term human pregnancy: effects of the oxytocin antagonist atosiban. Am J Obstet Gynecol. 1994 Dec;171(6):1634-42. doi: 10.1016/0002-9378(94)90415-4. PMID 7802081
- [Background] Mishra V, Agarwal H, Goel S, Roy P, Choudhary S, Lamba S. A Prospective Case-control Trial to Evaluate and Compare the Efficacy and Safety of Atosiban versus Placebo in In vitro Fertilization-embryo Transfer Program. J Hum Reprod Sci. 2018 Apr-Jun;11(2):155-160. doi: 10.4103/jhrs.JHRS_7_17. PMID 30158812
- [Background] Kimura T, Tanizawa O, Mori K, Brownstein MJ, Okayama H. Structure and expression of a human oxytocin receptor. Nature. 1992 Apr 9;356(6369):526-9. doi: 10.1038/356526a0. PMID 1313946
- [Background] Fanchin R, Righini C, Olivennes F, Taylor S, de Ziegler D, Frydman R. Uterine contractions at the time of embryo transfer alter pregnancy rates after in-vitro fertilization. Hum Reprod. 1998 Jul;13(7):1968-74. doi: 10.1093/humrep/13.7.1968. PMID 9740459
- [Background] Lan VT, Khang VN, Nhu GH, Tuong HM. Atosiban improves implantation and pregnancy rates in patients with repeated implantation failure. Reprod Biomed Online. 2012 Sep;25(3):254-60. doi: 10.1016/j.rbmo.2012.05.014. Epub 2012 Jun 16. PMID 22818095
- [Derived] Craciunas L, Tsampras N, Kollmann M, Raine-Fenning N, Choudhary M. Oxytocin antagonists for assisted reproduction. Cochrane Database Syst Rev. 2021 Sep 1;9(9):CD012375. doi: 10.1002/14651858.CD012375.pub2. PMID 34467530